CLINICAL TRIAL: NCT03247959
Title: Effectiveness of Active and Passive Distraction Techniques on Reducing Fear and Anxiety and Improving Oral Health Knowledge of Children Undergoing Extraction in the Dental Operatory - A Randomized Controlled Trial
Brief Title: Effectiveness of Active and Passive Distraction Techniques on Reducing Fear and Anxiety and Improving Oral Health Knowledge of Children Undergoing Extraction in the Dental Operatory- A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indira Gandhi Institute of Dental Science (Other)
Responsible Party: Principal Investigator, Swarna Kannan, Principal investigator, Indira Gandhi Institute of Dental Science
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGIDSIRB2016NDP27PGSKPPD
Record Dates: First submitted 2017-07-31; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Fear Anxiety
Keywords: oral health education, distraction, videogame

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A: Videogame distraction during extraction procedure
  Interventions: Behavioral: Video game distraction and video distraction
- Group B (Experimental): Group B: Video distraction during extraction procedure
  Interventions: Behavioral: Video game distraction and video distraction
- Group C (Active Comparator): group C: Verbatim during extraction procedure
  Interventions: Behavioral: Video game distraction and video distraction

INTERVENTIONS:
Behavioral: Video game distraction and video distraction — video game distraction and video distraction will be advocated during the extraction procedure

SUMMARY:
The Purpose of this study is to evaluate the effectiveness of active ( video game) and passive (video) distraction techniques on reducing fear and anxiety and improving oral health knowledge of children undergoing extraction in the dental operatory

DETAILED DESCRIPTION:
Dentists are expected to identify and effectively treat childhood dental diseases that are within the knowledge and skills acquired during their dental education. As every child is different, safe and effective treatment of oral diseases often requires modifying the child's behavior. Behavior guidance involves interaction of the dentist and dental team, the patient and the parent directed towards communication and education. Its goal is to ease fear and anxiety while promoting an understanding of the need for good oral health.

In 1936, Freud defined Anxiety as an unpleasant affective state or condition, which is characterized by all that is covered by the word 'nervousness' and it can be prevented by the avoidance of negative experiences and promotion of positive experiences in children attending the dental operatory.

In Pediatric dentistry, communicative management and appropriate use of commands have been used in both cooperative and uncooperative child.Commonly used techniques associated with this guiding process are tell-show-do, voice control, nonverbal communication, positive reinforcement and physical restraints. Even though these techniques decrease the perception of unpleasantness, avert negative behaviours, gain or maintain the patient's attention and compliance, it is impossible for pediatric dentists to divert their attention from perceiving pain during invasive dental procedures.

American Academy of Pediatric Dentistry (2008) described distraction as a technique of diverting the patient's attention from what may be perceived as an unpleasant procedure. According to McCaul and Malott, one must attend to the pain stimulus in order to perceive it and also experience the associated distress. Thus distraction might help in reducing the pain perception. As the individual's attentional capacity is finite, a distracting task that requires a great deal of the person's attentional resources should leave little attentional capacity available for processing painful stimuli.

Thus, highly engaging and interactive distraction activities that involve multiple sensory systems are likely to be more effective than more passive distractors or distracters that involve only one or two sensory systems. A number of recent distraction interventions for acute pain in children and adolescents have employed virtual reality (VR) technology in conjunction with either a passive distraction stimulus, such as a movie (Sullivan, Schneider, Musselman, Dummett, & Gardiner, 2000), or an interactive distraction activity, such as a computer game (Dahlquist et al., 2007). However, the actual benefit of VR technology over and above the benefits of the distracting stimulus that is experienced through the VR equipment has not been adequately tested in children.

It is observed from the literature review that only few studies were found on virtual reality distraction and their findings suggest that virtual reality can enhance the effects of distraction for some children and thus demands further research.

Dental problems in children occur due to their poor oral health knowledge and difficulty of parents in implementing healthy oral habits for their children at home. Thus in order to promote oral health knowledge, method of delivering it should be effective. Till date only one study has focused on educating oral health through video game, thus investigators planned this study on videogames as videogames has got extreme potential and is a favourite time pass for children nowadays. The videogame/ video are the interactive tools which would help educate children in a playful way. Hence this study is planned to compare three behaviour guiding techniques (active distraction using videogames, passive distraction using video and verbatim (verbal distraction) in children( participants) for guiding their behavior during dental procedure in a dental operatory. All these three techniques utilize instructions related to oral health. In addition to that, investigators have planned to assess whether these distraction techniques could effectively deliver Oral Health Education to children ( participants).

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 6-12yrs
2. Children requiring simple extraction ( Primary teeth with preshedding mobility)
3. Children requiring Infiltration LA only

Exclusion Criteria:

1. Children below 6 yrs and above 12 yrs
2. Children with special health care needs
3. Children requiring complicated extraction

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in fear during the treatment | 30 minutes
  Fear will be assessed before, during and after the treatment by assessing the participants pulse rate
Reduction in anxiety during the treatment | 30 minutes
  Anxiety will be assessed by using chotta-bheem chutki anxiety scale before, during and after the treatment

SECONDARY OUTCOMES:
Improvement in Oral health knowledge | 1 week
  oral health education related questionnaire will be given to the participants before the treatment to assess the baseline measure and knowledge will be assessed again after 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Swarna Kannan, Postgraduate, Principal Investigator — Indira gandhi institute of dental sciences
Locations (1):
- Swarna, Puducherry, Puducherry, India

IPD SHARING:
Plan to Share IPD: Undecided